CLINICAL TRIAL: NCT06853626
Title: Improved Management of Acute Chest Pain in Emergency Primary Care. The OUT-POC Study (One-hoUr Troponin Using a High-sensitivity Point-Of-Care Assay in Emergency Primary Care)
Brief Title: One-hoUr Troponin Using a High-sensitivity Point-Of-Care Assay in Emergency Primary Care
Acronym: OUT-POC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Health Association (Other); Oslo University Hospital (Other); QuidelOrtho (Industry); Vestre Viken Hospital Trust (Other); The Dam Foundation (Other); Amsterdam UMC (Other); Sørlandet Hospital (Unknown)
Responsible Party: Principal Investigator, Tonje R. Johannessen, Principal Investigator, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDAM_FOR555568
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction (AMI); Chest Pain; Acute Coronary Syndromes (ACS); Non-cardiac Chest Pain; Troponin; Point of Care Testing; Out-of-hours Medical Care; Primary Care
Keywords: TriageTrue; POC; hs-cTnI; 0/1-hour algorithm; troponin; chest pain; primary care; OOH; out-of-hours; acute myocardial infarction; point-of-care; OUT-POC; QuidelOrtho
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, investigator-initiated pre-post intervention study aiming to evaluate implementation of the QuidelOrthos TriageTrue hs-cTnI whole-blood assay at six Norwegian (non-randomised) emergency primary care clinics.
  A control group will be identified to estimate the effect of the OUT-POC protocol. We will benefit from registry data to 1) estimate hospital referrals before the intervention in the same regions and 2) establish an external control group consisting of municipalities that are not using POC hs-cTn testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TriageTrue hs-cTnI 0/1-hour algorithm (Other): Study participants will have a venous blood sample done for hs-cTnI testing using the QuidelOrthos TriageTrue whole-blood POC assay. The treating physician will evaluate the results using an assay-specific 0/1-hour algorithm (developed by Boeddinghaus et al., 2020).
  Interventions: Diagnostic Test: QuidelOrthos TriageTrue hs-cTnI whole-blood assay

INTERVENTIONS:
Diagnostic Test: QuidelOrthos TriageTrue hs-cTnI whole-blood assay — Already described

SUMMARY:
Acute chest pain is a prevalent medical emergency in primary emergency care settings. Triage of chest pain prior to hospital admission presents significant challenges due to the absence of sufficiently sensitive diagnostic tools. Clinical signs, symptoms, risk assessment scores, or a normal electrocardiogram (ECG) can reliably exclude acute myocardial infarction (MI). This diagnostic uncertainty has resulted in chest pain being the second most common cause for acute hospital referrals from Norwegian emergency primary care, even though chest pain is frequently non-cardiac in origin.

In acute MI events, cardiac troponins are released into the bloodstream from the damaged myocardium, where low values are used to exclude MI. Until recently, such testing has necessitated using high-sensitivity cardiac troponin (hs-cTn) assays, which have been limited to hospital laboratories. However, recent technological advancements in point-of-care (POC) testing allow access to whole-blood assays that meet high-sensitivity criteria.

In this upcoming project, the investigators will evaluate the implementation of a whole-blood POC assay (QuidelOrtho TriageTrue hs-cTnI) across six Norwegian emergency primary care clinics. The study plans to enrol 2,500 patients over a period of 1.5 years. The clinical performance of the novel strategy will be investigated, as well as its impact on healthcare utilization and hospital referrals compared to standard care. Additionally, the investigators will assess the prevalence of persistent chest pain and its effects on quality of life, alongside psychological stress and anxiety, through validated questionnaires.

This project aims to offer better and more comprehensive management of the large group of emergency primary care patients with acute chest pain, contributing to reduced hospital referrals, improved quality of life, and more sustainable use of healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18+ years) with non-traumatic acute chest pain presenting in emergency primary care
* Troponin testing requested by the treating physician

Exclusion Criteria:

* Acute STEMI (direct hospital referral required)
* Haemodynamically unstable (direct hospital referral required)
* Not able to provide written, informed consent (i.e., due to time restraints, language barriers, impaired cognitive function, or other reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of acute myocardial infarctions at the index episode | From baseline to 30 days
  Proportion of acute myocardial infarction at baseline, to assess the predictive performance of the TriageTrue 0/1-hour algorithm (incl. safety and accuracy) at index
PROM: Health-related quality of life | At baseline and repeated after 90 days
  Differences in health-related quality of life among chest pain participants will be assessed through self-reported EQ-5D questionnaire with five levels (EQ-5D-5L) incl. the EQ-5D visual analogue scale (EQ VAS).

SECONDARY OUTCOMES:
Efficiency | Baseline
  The proportion of patients finished triaged as rule-out or rule-in by the protocol at index
Total number of hospital referrals at index | Baseline
  Proportion of patients being directly hospitalised at index
Total length of stay | Baseline to 24 hours
  Total duration of the chest pain assessment at the clinic at index (i.e., time from arrival to discharge)
Composite of acute MI and all-cause death | From baseline to 1 year
  To assess the prognostic performance of the algorithm after 30, 90, and 365 days
PROM: Cardiac Anxiety | At baseline and repeated after 90 days
  Changes in cardiac-related anxiety, measured by the Cardiac Anxiety Questionnaire (CAQ)
PROM: Depression | At baseline and repeated after 90 days
  Changes in depression, measured by the Patient Health Questionnaire-4 (PHQ-4)
PROM: Insomnia | At baseline and repeated after 90 days
  Changes in sleep disturbances, measured by the Sleep Condition Indicator-02
PROM: Burden of chest pain | At baseline and repeated after 90 days
  Changes in chest pain frequency, avoidance, intensity and duration, measured by Jonsbu's questionnaire
Incremental cost-effectiveness ratio | From baseline to 1 year
  Difference in quality-adjusted life-years by using the OUT-POC protocol compared to standard care (control)
Societal costs | From baseline to 1 year
  Proportion of production loss/sick leave due to chest pain-related diagnoses
Healthcare utilization | From baseline to 1 year
  Total number and type of treatment and follow-up in primary and secondary care due to chest pain-related diagnoses
Healthcare costs | From baseline to 1 year
  Total costs of assessing patients with chest pain in emergency primary care by using the protocol compared to usual care (control), including unit costs per treatment, visit, stay.

OTHER OUTCOMES:
Performance of the TriageTrue hs-cTnI whole-blood assay and clinical risk scores | From baseline to 1 year
  Pre-planned subanalyses to evaluate the performance of various clinical risk scores integrating a single hs-cTnI POC measurement (incl. the History, Electrocardiogram, Age, Risk factors, and Troponin (HEART) score and the Troponin-only Manchester Acute Coronary Symdrome (T-MACS) score).

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - Lyngen Emergency Primary Care Centre, Lyngseidet, Lyngen
  - Alta Emergency Primary Care Centre, Alta
  - Drammen Emergency Primary Care Centre, Drammen
  - Fredrikstad and Hvaler Emergency Primary Care Centre, Fredrikstad
  - Oslo Accident and Emergency Outpatient Clinic, Oslo
  - Trondheim Intermunicipal Emergency Primary Care Centre, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johannessen TR, Vallersnes OM, Larstorp ACK, Halvorsen S, Atar D. One-Hour Troponin Using a High-Sensitivity Point-of-Care Assay in Emergency Primary Care: The OUT-POC Pilot Study. Cardiology. 2025 Mar 7:1-13. doi: 10.1159/000545127. Online ahead of print. PMID 40058362
- [Result] Johannessen TR, Vallersnes OM, Larstorp ACK, Halvorsen S, Atar D. Authors' Response Letter - Expanding the Use of Point-of-Care hs-cTnI in Emergency Primary Care: Insights from the OUT-POC Pilot Study. Cardiology. 2025 May 22:1-3. doi: 10.1159/000546344. Online ahead of print. No abstract available. PMID 40418919
- See also: OUT-POC pilot study — http://karger.com/crd/article/doi/10.1159/000546344/927465/Expanding-the-Use-of-Point-of-Care-hs-cTnI-in
- See also: OUT-POC pilot study; Authors' Response Letter — http://karger.com/crd/article/doi/10.1159/000545127/923307/One-Hour-Troponin-Using-a-High-Sensitivity-Point